CLINICAL TRIAL: NCT05696431
Title: Comparative Evaluation of Two-Year Clinical Performance of Three Universal Adhesives in Posterior Restorations
Brief Title: Clinical Performance of Three Universal Adhesives in Posterior Restorations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: A01041022
Record Dates: First submitted 2023-01-07; First posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-11

CONDITIONS: Recurrent Caries

STUDY DESIGN:
Intervention Model Description: Each patient will receive the three universal adhesives with the same restorative material randomly in three posterior teeth. All the materials will be used according to their manufacturers' instructions.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Universal adhesive (Placebo Comparator): After preparation of three posterior cavities in each patient. The cavities will be randomly divided into three groups according to the type of the adhesive used. This group will receive a universal adhesive as control group.
  Interventions: Other: Universal adhesives application
- Fluoride-releasing universal adhesive (Active Comparator): After preparation of three posterior cavities in each patient. The cavities will be randomly divided into three groups according to the type of the adhesive used. This group will receive a Fluoride-releasing universal adhesive.
  Interventions: Other: Fluoride-releasing universal adhesive
- Universal adhesive with bioactive properties (Active Comparator): After preparation of three posterior cavities in each patient. The cavities will be randomly divided into three groups according to the type of the adhesive used.This group will receive a universal adhesive with bioactive properties.
  Interventions: Other: universal adhesive with bioactive properties

INTERVENTIONS:
Other: Universal adhesives application — The adhesive will be used according to their manufacturer's instructions. Selective etching for enamel will be applied for 15 seconds, followed by rinsing and gentle air drying. Then, the adhesive will be applied to enamel and dentin and light cured using a light-curing unit for 20 seconds. The composite material will be incrementally applied, and each increment will be light cured for 20 seconds. The restoration will be finished and polished using finishing and polishing instruments.
  Arms: Universal adhesive
Other: universal adhesive with bioactive properties — The adhesive will be used according to their manufacturer's instructions. Enamel and dentin will be cleaned using clean and boost for 10 seconds, rinsed and gently dried. Then, the adhesive will be applied to enamel and dentin and light cured using a light-curing unit for 20 seconds. The composite material will be incrementally applied, and each increment will be light cured for 20 seconds. The restoration will be finished and polished using finishing and polishing instruments.
  Arms: Universal adhesive with bioactive properties
Other: Fluoride-releasing universal adhesive — Fluoride-releasing universal adhesive
  Arms: Fluoride-releasing universal adhesive

SUMMARY:
This study was designed to evaluate and compare the two-year clinical performance of three universal adhesives in posterior composite restorations, based on International dental federation (FDI) criteria.

DETAILED DESCRIPTION:
The description of the experimental design will follow the Consolidated Standards of Reporting Trials (CONSORT) statement. The present study will be a double blinded (patients and examiner) randomized clinical trial anticipating the split-mouth design. 30 adult patients seeking dental treatment in Operative Department clinic at Faculty of Dentistry, Mansoura University will be enrolled in the current study with a total of 90 teeth with Class I or II posterior composite restorations.

No advertisement will be made for participant recruitment, forming a sample of convenience. Each patient will sign a consent form before participating in the current study. The study will be conducted from November 2022 to November 2024 as a part of Doctoral dissertation. Mansoura University institution's ethics committee approved the form and protocol before conducting the study. The sample size was calculated based on a previous study with a similar study design. Parameters including a significance level of 5% (p < 0.05) and a power of 80% were used to calculate an appropriate sample size of 28 cases. Allowing for a 20% drop-out rate, the total sample size was set at 30 cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients will have at least 3 posterior teeth with carious lesions of ICDAS score 4, or 5.
* The teeth will have to be vital, without spontaneous pain and/or mobility.
* Patients must have a good oral hygiene.
* Patients with normal and full occlusion.

Exclusion Criteria:

* High caries risk patients with extremely poor oral hygiene.
* Patients with abutments.
* Patients with heavy bruxism habits and clenching.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-05 (Actual); Primary Completion 2024-11-05 (Estimated); Study Completion 2024-11-05 (Estimated)

PRIMARY OUTCOMES:
Aesthetic, functional and biological properties for composite restorations | 2 years after restorations application
  Composite restorations will be clinically assessed based on International dental federation (FDI) criteria.
  Scores from 1 to 5,
  1. Clinically excellent
  2. Clinically good
  3. Clinically sufficient
  4. Clinically unsatisfactory
  5. Clinically poor

SECONDARY OUTCOMES:
Radiographic examination | 2 years after restorations application
  Restorative materials will be examined radiographically every 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Yassmine F El-Sayed, Assis.Lec, Principal Investigator — Faculty of Dentistry, Mansoura University
Locations (1):
- Faculty of dentistry-Mansoura university, Al Mansurah, Dakahia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available within 6 Months for 2 years